CLINICAL TRIAL: NCT03135665
Title: Using Radiation-free Ultrasound for Screening Scoliosis Among School Children in Hong Kong to Reduce Unnecessary X-ray Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz-ping Lam, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ScoE_Protocol_V04
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ScoE (Other): This is a cross-sectional study on screened school children recommended for radiographic assessment in the scoliosis screening program of SHS in Hong Kong. Both x-ray, ultrasound and ATR measurement of the spine will be performed on the same day at Prince of Wales Hospital.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Scolioscan, the ultrasound system reported to be reliable and valid for spinal deformity assessment, will be used. The system composes of an ultrasound scanner with a linear probe of 100 mm in width and frequency range of 4-10MHz, a frame structure and a spatial sensor which is attached to the ultrasound probe for spatial data capture. Daily calibration will be performed using a phantom to assure accuracy of spine image formation and subsequent angle measurement.
  Subjects will stand on the Scolioscan platform with a standardized posture kept stable with pegs throughout the scanning process.. After adjusting the ultrasound scanner setting, the probe will be steered from L5 to T1 spinous process for scanning.
  SPA will be used to determine the ultrasound-based Referral Status through predicting whether the Cobb angle is beyond the referral threshold of ≥20° or not. There are two values for the Referral Status: either "for specialist referral" or "not for specialist referral".
  Other Names: Scolioscan

SUMMARY:
In the scoliosis screening program of the Student Health Service (SHS), Department of Health (DH), in Hong Kong, more than 50% of screened school children prescribed with x-ray examination basing on the screening protocol did not have Cobb angle greater than the referral threshold of 20°; ie they did not need specialist referral and thus were subjected to unnecessary x-ray exposure. Our primary objective is to determine whether a new radiation-free ultrasound system could identify subjects with Cobb angle greater than the referral threshold of 20° thus avoiding unnecessary x-rays in the referral workflow. The secondary objective is to evaluate if Angle of Trunk Rotation (ATR) can further increase the accuracy of ultrasound assessment.

ELIGIBILITY:
Inclusion Criteria:

i. Schoolchildren in Hong Kong attending School Screening Program provided by Student Health Service ii. Recommended for radiographic assessment in the scoliosis screening program

Exclusion Criteria:

* i. Patients with standing height <1 m, or >2 m ii. Patients with body mass index (BMI) ≥25 kg/m2 iii. Subjects with skin diseases iv. Subjects with fracture or wound that affect ultrasound scanning v. Subjects with ferromagnetic implants vi. Subjects with surgery done for the spine vii. Subjects with winged scapula or other irregularity of back contour that affect ultrasound scanning viii. Subjects who cannot stand steadily during scanning ix. Subjects with allergy to ultrasound gel

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 442 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
ultrasound-based Referral Status | Baseline
  "for specialist referral" or "not for specialist referral", through predicting whether the Cobb angle is beyond the referral threshold of ≥20° or not in scoliosis screening

SECONDARY OUTCOMES:
ATR | Baseline
  evaluate if this parameter can increase the accuracy of ultrasound assessment

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ping Lam, Principal Investigator — Assistant Professor (Clinical)
Locations (1):
- Department of Orthopaedics and Traumatology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] COBB JR. The problem of the primary curve. J Bone Joint Surg Am. 1960 Dec;42-A:1413-25. No abstract available. PMID 14448728
- [Background] Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Effects of bracing in adolescents with idiopathic scoliosis. N Engl J Med. 2013 Oct 17;369(16):1512-21. doi: 10.1056/NEJMoa1307337. Epub 2013 Sep 19. PMID 24047455
- [Background] Hresko MT, Talwalkar V, Schwend R; AAOS, SRS, and POSNA. Early Detection of Idiopathic Scoliosis in Adolescents. J Bone Joint Surg Am. 2016 Aug 17;98(16):e67. doi: 10.2106/JBJS.16.00224. No abstract available. PMID 27535448
- [Background] Luk KD, Lee CF, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Fong DY. Clinical effectiveness of school screening for adolescent idiopathic scoliosis: a large population-based retrospective cohort study. Spine (Phila Pa 1976). 2010 Aug 1;35(17):1607-14. doi: 10.1097/BRS.0b013e3181c7cb8c. PMID 20453727
- [Background] Fong DY, Lee CF, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Luk KD. A meta-analysis of the clinical effectiveness of school scoliosis screening. Spine (Phila Pa 1976). 2010 May 1;35(10):1061-71. doi: 10.1097/BRS.0b013e3181bcc835. PMID 20393399
- [Background] Lee CF, Fong DY, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Luk KD. Costs of school scoliosis screening: a large, population-based study. Spine (Phila Pa 1976). 2010 Dec 15;35(26):2266-72. doi: 10.1097/BRS.0b013e3181cbcc10. PMID 20531070
- [Background] Lee CF, Fong DY, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Luk KD. Referral criteria for school scoliosis screening: assessment and recommendations based on a large longitudinally followed cohort. Spine (Phila Pa 1976). 2010 Dec 1;35(25):E1492-8. doi: 10.1097/BRS.0b013e3181ecf3fe. PMID 21102278
- [Background] Fong DY, Cheung KM, Wong YW, Wan YY, Lee CF, Lam TP, Cheng JC, Ng BK, Luk KD. A population-based cohort study of 394,401 children followed for 10 years exhibits sustained effectiveness of scoliosis screening. Spine J. 2015 May 1;15(5):825-33. doi: 10.1016/j.spinee.2015.01.019. Epub 2015 Jan 20. PMID 25615844
- [Background] Hoffman DA, Lonstein JE, Morin MM, Visscher W, Harris BS 3rd, Boice JD Jr. Breast cancer in women with scoliosis exposed to multiple diagnostic x rays. J Natl Cancer Inst. 1989 Sep 6;81(17):1307-12. doi: 10.1093/jnci/81.17.1307. PMID 2769783
- [Background] Doody MM, Lonstein JE, Stovall M, Hacker DG, Luckyanov N, Land CE. Breast cancer mortality after diagnostic radiography: findings from the U.S. Scoliosis Cohort Study. Spine (Phila Pa 1976). 2000 Aug 15;25(16):2052-63. doi: 10.1097/00007632-200008150-00009. PMID 10954636
- [Background] Schmitz-Feuerhake I, Pflugbeil S. 'Lifestyle' and cancer rates in former East and West Germany: the possible contribution of diagnostic radiation exposures. Radiat Prot Dosimetry. 2011 Sep;147(1-2):310-3. doi: 10.1093/rpd/ncr348. Epub 2011 Aug 10. PMID 21835840
- [Background] Suzuki S, Yamamuro T, Shikata J, Shimizu K, Iida H. Ultrasound measurement of vertebral rotation in idiopathic scoliosis. J Bone Joint Surg Br. 1989 Mar;71(2):252-5. doi: 10.1302/0301-620X.71B2.2647754.
- [Background] Huang QH, Zheng YP, Lu MH, Chi ZR. Development of a portable 3D ultrasound imaging system for musculoskeletal tissues. Ultrasonics. 2005 Jan;43(3):153-63. doi: 10.1016/j.ultras.2004.05.003. PMID 15556650
- [Background] Cheung CW, Law SY, Zheng YP. Development of 3-D ultrasound system for assessment of adolescent idiopathic scoliosis (AIS): and system validation. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:6474-7. doi: 10.1109/EMBC.2013.6611037. PMID 24111224
- [Background] Purnama KE, Wilkinson MH, Veldhuizen AG, van Ooijen PM, Lubbers J, Burgerhof JG, Sardjono TA, Verkerke GJ. A framework for human spine imaging using a freehand 3D ultrasound system. Technol Health Care. 2010;18(1):1-17. doi: 10.3233/THC-2010-0565. PMID 20231799
- [Background] Li M, Cheng J, Ying M, Ng B, Zheng YP, Lam TP, Wong WY, Wong MS. Could clinical ultrasound improve the fitting of spinal orthosis for the patients with AIS? Eur Spine J. 2012 Oct;21(10):1926-35. doi: 10.1007/s00586-012-2273-4. Epub 2012 Mar 25. PMID 22447408
- [Background] Chen W, Lou EH, Zhang PQ, Le LH, Hill D. Reliability of assessing the coronal curvature of children with scoliosis by using ultrasound images. J Child Orthop. 2013 Dec;7(6):521-9. doi: 10.1007/s11832-013-0539-y. Epub 2013 Oct 22. PMID 24432116
- [Background] Ungi T, King F, Kempston M, Keri Z, Lasso A, Mousavi P, Rudan J, Borschneck DP, Fichtinger G. Spinal curvature measurement by tracked ultrasound snapshots. Ultrasound Med Biol. 2014 Feb;40(2):447-54. doi: 10.1016/j.ultrasmedbio.2013.09.021. Epub 2013 Nov 19. PMID 24268452
- [Background] Li M, Cheng J, Ying M, Ng B, Lam TP, Wong MS. A Preliminary Study of Estimation of Cobb's Angle From the Spinous Process Angle Using a Clinical Ultrasound Method. Spine Deform. 2015 Sep;3(5):476-482. doi: 10.1016/j.jspd.2015.03.001. Epub 2015 Oct 2. PMID 27927534
- [Background] Cheung CW, Zhou GQ, Law SY, Mak TM, Lai KL, Zheng YP. Ultrasound Volume Projection Imaging for Assessment of Scoliosis. IEEE Trans Med Imaging. 2015 Aug;34(8):1760-8. doi: 10.1109/TMI.2015.2390233. Epub 2015 Jan 12. PMID 25594962
- [Background] Zheng YP, Lee TT, Lai KK, Yip BH, Zhou GQ, Jiang WW, Cheung JC, Wong MS, Ng BK, Cheng JC, Lam TP. A reliability and validity study for Scolioscan: a radiation-free scoliosis assessment system using 3D ultrasound imaging. Scoliosis Spinal Disord. 2016 May 31;11:13. doi: 10.1186/s13013-016-0074-y. eCollection 2016. PMID 27299162
- [Background] Morrison DG, Chan A, Hill D, Parent EC, Lou EH. Correlation between Cobb angle, spinous process angle (SPA) and apical vertebrae rotation (AVR) on posteroanterior radiographs in adolescent idiopathic scoliosis (AIS). Eur Spine J. 2015 Feb;24(2):306-12. doi: 10.1007/s00586-014-3684-1. Epub 2014 Nov 21. PMID 25412836
- [Background] Lowe T, Berven SH, Schwab FJ, Bridwell KH. The SRS classification for adult spinal deformity: building on the King/Moe and Lenke classification systems. Spine (Phila Pa 1976). 2006 Sep 1;31(19 Suppl):S119-25. doi: 10.1097/01.brs.0000232709.48446.be. PMID 16946628